CLINICAL TRIAL: NCT02170701
Title: Multicenter, Open-label, Ascending Dose Study of BIBR 1048 in the Prevention of Venous Thromboembolism in Patients Undergoing Primary Elective Total Hip Replacement Surgery. Bistro I
Brief Title: BIBR 1048 in the Prevention of Venous Thromboembolism in Patients Undergoing Primary Elective Total Hip Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.11
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (1):
- BIBR 1048 (Experimental): Ascending doses (in mg) given twice daily
  Interventions: Drug: BIBR 1048

INTERVENTIONS:
Drug: BIBR 1048 — Ascending doses (in mg) given twice daily

SUMMARY:
* To determine the therapeutic window of BIBR 1048 in order to select doses for further studies in the development plan.
* Twice daily regimen will be tested for most dose levels and once daily administration will also be evaluated when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a primary elective total hip replacement
* Male of female being 18 years or older
* Patients weighing at least 40 kg
* Written informed consent for study participation

Exclusion Criteria:

* Bleeding diathesis, constitutional or acquired coagulation disorders
* Major surgery or trauma (e.g. hip fracture) within the last three months. Patients with previous hip fractures associated with plate revisions at any time will be excluded
* Cardiovascular disease including uncontrolled hypertension at time of enrolment or history of myocardial infarction within the last 6 months
* Any history of haemorrhagic stroke, intracranial or intraocular bleeding or cerebral ischaemic attacks
* Known history of deep venous thrombosis (DVT)
* Gastrointestinal or pulmonary bleeding within the last year
* Known liver disease Aspartate transaminase (AST) or Alanine transaminase (ALT) > 3 x ULN)
* Known renal disease (serum creatinine > 1.5 x ULN)
* Use of long- term anticoagulants, antiplatelet drugs, or fibrinolytics within 7 days prior to hip replacement operation (also contraindicated during the period of prophylaxis)
* Women of childbearing potential
* Known allergy to radiopaque contrast media
* Known thrombocytopenia (prior platelet count below 100,000 cells/microliter)
* Active malignant disease
* Current H2 blocker or proton pump inhibitor treatment
* Current cytostatic treatment
* Treatment with an investigational drug in the past month
* Leg amputee
* Known alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2000-10; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Rate of venous thrombolic events | Up to day 10 after hip surgery
Changes from baseline in activated partial thromboplastin time (aPTT) | From baseline (day -14 to day -1 before treatment) until last day of treatment (up to day 10)
Changes from baseline in ecarin clotting time (ECT) | From baseline (day -14 to day -1 before treatment) until last day of treatment (up to day 10)
Changes from baseline in thrombin time (TT) | From baseline (day -14 to day -1 before treatment) until last day of treatment (up to day 10)
Rate of major bleeding events during treatment phase | Start of treatment (day 0) until end of treatment (up to day 10)
Cpre,ss (predose plasma concentrations at steady state) | baseline and predose from day 1 to last treatment day
Cmax,ss (maximum plasma concentration at steady state (day 4)) | Day 4
Tmax,ss (time to reach Cmax,ss) | baseline, day 0 before and 4 hours after, day 1 to 4 before and 2 h after treatment, day 5 to last treatment day before treatment
CLtot/f (total clearance of drug from plasma after oral administration) | baseline, day 0 before and 4 hours after, day 1 to 4 before and 2 h after treatment, day 5 to last treatment day before treatment
AUCss (area under the plasma concentration curve of one dosing interval at steady state) | baseline, day 0 before and 4 hours after, day 1 to 4 before and 2 h after treatment, day 5 to last treatment day before treatment
PTF (percent peak trough fluctuation for the last dosing interval) | baseline, day 0 before and 4 hours after, day 1 to 4 before and 2 h after treatment, day 5 to last treatment day before treatment
Cmax,ss (maximum plasma concentration at steady state (day 4)) | Day 4 before and 0.5, 1, 2, 4 , 8, 12 , 14 h after treatment

SECONDARY OUTCOMES:
Venous thromboembolism diagnosed during the follow-up period | Up to 6 weeks after surgery (day 42)